CLINICAL TRIAL: NCT06210464
Title: Disease and Biomarker Profiling of Chinese Lupus Nephritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nan Shen (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Nan Shen, Chief physician, RenJi Hospital
Organization: RenJi Hospital (Other)
Other Study IDs: BASICHR0060
Record Dates: First submitted 2023-12-18; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Characterize the Molecular Profile of Lupus Nephritis(LN) Patients to Understand Themechanism(s)Contributing to Patient Responsiveness to Soc; Integrated Analysis of LN Patient Molecular Profiling and Clinical Annotations to Understand LNdisease Heterogeneity for Disease Endotype; Validate the Association of the Candidate Biomarker Panel Proposed in Table 3-1 With LN Diseasemonitoring

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — Trial have no Intervention measures.

SUMMARY:
In the proposed study , Novartis Institutes of Biomedical Research ( NIBR ) collaborates with Reni HospitalAffiated to Shanghai Jiaotong University School of Medicine ( Ren ) , aiming to identify particular LNendotype , and to discover novel biomarkers which link the endotype to disease phenotype , especially todisease monitorng , treatment response and prognosis prediction . The study proposes to take bothcandidate approach ( reported biomarkers ) and unbiased high-throughput proteomics profiling tools( Somascan measures up to 7,000 protein analytes ) to analyze 100 Class I / V LN patients with welldocumented clinical annotation , treatment schedule and disease follow up . Both serum / plasma and urrpatients will be extensively characterized with a focus on non-invasive biomarkediscovery and validation . Integrated analysis will be performed to associate patient molecular signature withtheir clinical annotation , renal pathology features , and response to Soc treatment . We will generahypothesis from these analyses to propose molecular markers to predict patient response to Soc treatmentand to endotype the disease , discover the mechanisms that could contrbute to unsatisfactory response toSoc , and identity more specific and sensitive non-invasive biomarkers in serum or urine that can be used in disease monitoring , disease prognosis and patient stratificationproposed study Will help usunderstand the heterogeneity of LN at the molecular level , which could be an essential first step towardsLN precision medicine . It will provide scientific rationale for improved LN clinical diagnosis , novel therapeutichypothesis , patient stratification , clinical study design and combination strategy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to communicate well with investigator, understand the study procedures and provide writteninformed consent before any study-related sample/data are accesse 2. Men and women with systemic lupus erythematosus (see below), aged 18 years and 75 years fulfilling 1997 ACR classification criteria for SLE, or 2012 SLICC classification criteria for SLE,OI2020 eularacr classification criteria for sstological diagnosis of proliferative lupusnephritis wealth OrganizationO)ISN/RPS (Weening et al 2004) Class I or class IV,with soc treatment anddisease monitoringleast one year 3. Serum/plasma and urine samples were collected at baseline of the treatme

Exclusion Criteria:

* 1.Presence of another autoimmune rheumatic disease that is active and constitutes the principalIllness , except for rheumatoid arthritis , Sjogrens syndrome and autoimmune thyroiditis 2 . Any glomerulonephritis other than WHO Class l or V lupus nephritis Patients with proliferativenephritis ( Class l or V ) who , in addition , have overlapping histological signs for other glomerulonephritis , e.g. , Class V are eligible at the investigator s discretion 3. History of malignancy with the exception of basal cell or squamous cell carcinoma of the skin orsitu carcinoma of the cervix within the last 2 vears 4 . Urinary system infection 5 . Pregnant women

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: aged 18 years and 75 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-14 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Serum SDMA : serum EMIT or LC-MS assayUrinary | 2025
SCD163 : urine ELISA assay | 2025
Urine RALL Index ( NGAL , KIM-1 , MCP-1 , Adiponectin , Ceruloplasmin andHemopexin ) 4-plex panel ELLA and two single-plex ELISA | 2025
Urine Creatinine urine BM data normalization , enzymatic method on Cobas | 2025